CLINICAL TRIAL: NCT06620406
Title: Pilot Study of Synbiotic Therapy for Neuropsychiatric PASC
Brief Title: Synbiotic Therapy for NP-PASC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Michael Yin, Associate Professor of Medicine, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AAAV3630
Record Dates: First submitted 2024-09-26; First posted 2024-10-01 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Post-Acute COVID-19 Syndrome; Long COVID-19
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Synbiotic Therapy (Experimental): A mixture of the prebiotic potato resistant starch (RS, Bobs Red Mill) and the probiotic IVS-1 (Bifidobacterium adolescentis).
  Interventions: Dietary Supplement: Synbiotic IVS-1
- Placebo (Placebo Comparator): The placebo to be used is Maltodextrin, a carbohydrate packaged similarly to the study intervention.
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Synbiotic IVS-1 — A mixture of the prebiotic potato resistant starch (RS, Bobs Red Mill) and the probiotic IVS-1 (Bifidobacterium adolescentis).
  Other Names: Prebiotic+Probiotic
  Arms: Synbiotic Therapy
Dietary Supplement: Maltodextrin — Maltodextrin, a carbohydrate packaged similarly to the study intervention
  Arms: Placebo

SUMMARY:
Gut microbiome dysbiosis has been noted in patients with Post-acute sequelae (PASC) of Severe Acute Respiratory Syndrome-CoronaVirus -2 (SARS-CoV-2). A study performed at Columbia found that plasma levels of the short chain fatty acid (SCFA), butyric acid, remained lower in people with Neuropsychiatric PASC (NP-PASC) than in people with PASC after SAR-CoV-2 infection. Synbiotics improve SCFA levels and are well-tolerated in the general population but have not been studied among people with PASC in the United States. The purpose of this pilot study is to characterize changes in plasma SCFA levels and gut microbiome after treatment with synbiotics and placebo in people with NP-PASC. The intervention will be a mixture of the prebiotic resistant starch and the probiotic Bifidobacterium adolescentis in-vivo selection 1 strain (iVS-1). The placebo will be Maltodextrin.

DETAILED DESCRIPTION:
In this pilot study, up to 30 participants with NP-PASC at Columbia University Medical Center (CUIMC) will be randomized to take the intervention (n=15) or placebo (n=15). Both intervention and placebo will be similar in terms of appearance and taste, and participants will be asked to take the intervention or placebo with water twice daily, for up to 4 weeks. At the enrollment and study follow-up visit, the investigators will obtain data on acceptability and feasibility, including feasibility of assessing adherence and outcomes, and collect blood, rectal swabs and stool for outcome assessment.

The study intervention is a mixture of the prebiotic potato RS (Bobs Red Mill) and the probiotic IVS-1 (Bifidobacterium adolescentis). One dose will be RS and IVS-1 mixed together in a single-use sachet. The placebo will be Maltodextrin, a carbohydrate, packaged similarly to the intervention. Participants will take one dose twice daily with water, for 4 weeks. Each participant will receive a 4-week supply of sachets at the screening/enrollment visit.

There will be a total of two visits: screening/enrollment/randomization and week 4. During the screening visit, study information will be provided to potential participants, and interested participants will sign an informed consent and undergo screening procedures. Those who meet eligibility criteria will then undergo enrollment and randomization procedures on the same day. Data on sociodemographic and medical history will be collected using surveys, and relevant samples will also be collected at the first visit as well as a self-administered rectal swab, and self-collected stool for gut microbiome studies and blood test for SCFA levels. The participant will then initiate the intervention or placebo, and the study staff will counsel and support the participants on administration of the intervention or placebo. At the 4-week visit, clinical data and samples will be collected, as well as data on acceptability, feasibility, adherence.

ELIGIBILITY:
Inclusion Criteria:

1. >18 years of age,
2. Prior mild acute SARS-CoV-2 infection (positive testing by FDA approved antigen or molecular test or positive anti-nucleocapsid antibody) and not requiring hospitalization
3. Meeting Center for Disease Control (CDC) criteria for PASC (any new or recurrent symptom present >4 weeks after SARS-COV-2 infection)
4. Meeting 2015 Institute of Medicine (IOM) criteria for myalgic encephalomyelitis/chronic fatigue syndrome (ME-CFS) of 3 required symptoms for fatigue to select for individuals specifically with NP-PASC (a substantial reduction or impairment in ability to engage in pre-illness levels of activity, post-exertional malaise, and unrefreshing sleep) and at least one of the two following manifestations (cognitive impairment or orthostatic intolerance).
5. meets cognitive impairment threshold on neurocognitive battery.

Exclusion Criteria:

1. Pregnancy or breastfeeding
2. Currently taking or using the following non-study products within 30 days prior to study entry:

   * probiotics, prebiotics, or fiber supplements
   * immunosuppressive or immunomodulatory drugs
   * antibiotics
3. Heavy drug or alcohol use
4. Known allergy to any of the study products
5. Serious illness requiring systemic treatment and/or hospitalization within 30 prior to study entry
6. Liver cirrhosis, history of inflammatory bowel disease, or other major conditions related to colon
7. Any episode of acute or persistent diarrhea within 1 day prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2024-12-09 (Actual); Primary Completion 2025-08-06 (Actual); Study Completion 2025-08-06 (Actual)

PRIMARY OUTCOMES:
Difference in plasma short chain fatty acid (SCFA) levels between study arms | 4 weeks
  SCFA levels will be measured from plasma samples and compared between the intervention group and the placebo group. In-group differences will also be measured between baseline and 4 weeks.
Difference in gut microbiota between study arms | 4 weeks
  Bacterial flora will be measured from rectal swab samples and compared between the intervention group and the placebo group. In-group differences will also be measured between baseline and 4 weeks.
Difference in other biomarkers between study arms | 4 weeks
  Additional biomarkers, such as serotonin and inflammatory cytokines, measured from the plasma samples and rectal swabs, whose concentration will be compared between the intervention group and the placebo group, and in-group differences between timepoints. Additional biomarkers include, but are not limited to, inflammatory cytokines and serotonin.
Difference in clinical profiles between study arms | 4 weeks
  Survey data will be compared between the intervention group and the placebo group, and in-group differences between timepoints. Survey data includes, but is not limited to, medication, COVID History, Vaccine History, and Medical History.

SECONDARY OUTCOMES:
Number of participants enrolled per week and agree to take the intervention | 4 weeks
  This measures the feasibility and acceptability of the study drug.
Number of participants who successfully take the intervention | 4 weeks
  This measures the feasibility and acceptability of the study drug.
Difference in NP-PASC symptoms between study arms | 4 weeks
  NP-PASC symptom severity differences as assessed by the NeuroScreen app between the baseline and the 4 week timepoint, and differences between the intervention and the placebo group.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Yin, MD, MS, Principal Investigator — Columbia University; Rupak Shivakoti, PhD, MHS, Principal Investigator — Columbia Universtiy Medical Center
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Participant confidentiality will be maintained and individual participant data will not be provided to other researchers, and there is no plan to do so.

REFERENCES:
- [Background] Liu Q, Mak JWY, Su Q, Yeoh YK, Lui GC, Ng SSS, Zhang F, Li AYL, Lu W, Hui DS, Chan PK, Chan FKL, Ng SC. Gut microbiota dynamics in a prospective cohort of patients with post-acute COVID-19 syndrome. Gut. 2022 Mar;71(3):544-552. doi: 10.1136/gutjnl-2021-325989. Epub 2022 Jan 26. PMID 35082169
- [Background] Kearney SM, Gibbons SM, Erdman SE, Alm EJ. Orthogonal Dietary Niche Enables Reversible Engraftment of a Gut Bacterial Commensal. Cell Rep. 2018 Aug 14;24(7):1842-1851. doi: 10.1016/j.celrep.2018.07.032. PMID 30110640
- [Background] Pandey KR, Naik SR, Vakil BV. Probiotics, prebiotics and synbiotics- a review. J Food Sci Technol. 2015 Dec;52(12):7577-87. doi: 10.1007/s13197-015-1921-1. Epub 2015 Jul 22. PMID 26604335
- [Background] Maldonado-Gomez MX, Martinez I, Bottacini F, O'Callaghan A, Ventura M, van Sinderen D, Hillmann B, Vangay P, Knights D, Hutkins RW, Walter J. Stable Engraftment of Bifidobacterium longum AH1206 in the Human Gut Depends on Individualized Features of the Resident Microbiome. Cell Host Microbe. 2016 Oct 12;20(4):515-526. doi: 10.1016/j.chom.2016.09.001. Epub 2016 Sep 29. PMID 27693307
- [Background] Sonnenburg ED, Smits SA, Tikhonov M, Higginbottom SK, Wingreen NS, Sonnenburg JL. Diet-induced extinctions in the gut microbiota compound over generations. Nature. 2016 Jan 14;529(7585):212-5. doi: 10.1038/nature16504. PMID 26762459
- [Background] Committee on the Diagnostic Criteria for Myalgic Encephalomyelitis/Chronic Fatigue Syndrome; Board on the Health of Select Populations; Institute of Medicine. Beyond Myalgic Encephalomyelitis/Chronic Fatigue Syndrome: Redefining an Illness. Washington (DC): National Academies Press (US); 2015 Feb 10. Available from http://www.ncbi.nlm.nih.gov/books/NBK274235/ PMID 25695122
- [Background] Grooms KN, Ommerborn MJ, Pham DQ, Djousse L, Clark CR. Dietary fiber intake and cardiometabolic risks among US adults, NHANES 1999-2010. Am J Med. 2013 Dec;126(12):1059-67.e1-4. doi: 10.1016/j.amjmed.2013.07.023. Epub 2013 Oct 15. PMID 24135514